CLINICAL TRIAL: NCT04862715
Title: Multicentre Prospective Double-blind Randomised Controlled Trial of the Effect of Intravenous Iron Supplementation and Exercise Training in Iron-deficient, But Not Anaemic, Patients With Chronic Kidney Disease on Exercise Capacity, Physical Function, Fatigue, and Skeletal Muscle Metabolism
Brief Title: The Iron and Muscle Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 234820
Record Dates: First submitted 2019-04-03; First posted 2021-04-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: CKD Stage 3; CKD Stage 4; Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Active study medication Medication name: Ferinject® Active ingredient: Ferric carboxymaltose Dosage form: 50 mg iron/ml solution for injection/infusion. Appearance: Dark brown, non-transparent aqueous solution Excipients: Sodium hydroxide, hydrochloric acid and water for injection Strength/Packaging: Each 2 ml vial contains 100 mg of iron as ferric carboxymaltose.
  Each 10 ml vial contains 500 mg of iron as ferric carboxymaltose. Each 20 ml vial contains 1,000 mg of iron as ferric carboxymaltose. Manufacturer: Vifor Pharma UK Limited
  Interventions: Drug: Ferinject
- Placebo (Placebo Comparator): Medication name: NaCl (sodium chloride 0.9%) Active ingredient: NaCl (sodium chloride 0.9%) Dosage form: 0.9% w/v NaCl as sterile solution in water for injection Excipients: Water Strength/Packaging: 100 ml container with 100 ml normal saline Manufacturer: As per local hospital supplier
  Interventions: Other: Placebo: NaCl (sodium chloride 0.9%)

INTERVENTIONS:
Drug: Ferinject — Active study medication Medication name: Ferinject® Active ingredient: Ferric carboxymaltose Dosage form: 50 mg iron/ml solution for injection/infusion. Appearance: Dark brown, non-transparent aqueous solution Excipients: Sodium hydroxide, hydrochloric acid and water for injection Strength/Packaging: Each 2 ml vial contains 100 mg of iron as ferric carboxymaltose.
  Each 10 ml vial contains 500 mg of iron as ferric carboxymaltose. Each 20 ml vial contains 1,000 mg of iron as ferric carboxymaltose. Manufacturer: Vifor Pharma UK Limited
  Arms: Treatment
Other: Placebo: NaCl (sodium chloride 0.9%) — Medication name: NaCl (sodium chloride 0.9%) Active ingredient: NaCl (sodium chloride 0.9%) Dosage form: 0.9% w/v NaCl as sterile solution in water for injection Excipients: Water Strength/Packaging: 100 ml container with 100 ml normal saline Manufacturer: As per local hospital supplier
  Arms: Placebo

SUMMARY:
This is a multi-center randomized controlled trial that will examine the efficacy of IV iron supplementation when compared to placebo, with and without exercise training, on changes in patient exercise capacity. The study aims to provide sufficient data to inform a power calculation for the definitive study to examine whether IV iron therapy in patients with CKD stages 3-4 (non-dialysis) can improve exercise capacity, muscle metabolism and physical function. Specifically, we propose to examine whether a strategy of IV iron therapy in patients with stages 3-4 CKD who are iron-deficient but NOT anaemic leads to improvements in exercise capacity.

Very little is currently known about the effects of iron deficiency on cardiac or skeletal muscle metabolism in patients suffering from CKD. Nevertheless, it seems likely that iron deficiency will contribute to mitochondrial dysfunction and reduced energy production in cardiac or skeletal muscle of CKD patients, and importantly may contribute to the reduced exercise capacity, physical function and overwhelming fatigue commonly reported in this population. The results of this trial will provide data to ascertain whether intravenous iron therapy might be beneficial to exercise capacity, muscle metabolism, physical function, and fatigue and whether iron repletion enhances the effect of an exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established CKD (Stages 3-4) not on dialysis
* Resting BP ≤ 160/95mmHg
* Men and women aged 18 - 80 years
* Serum ferritin level less than 100μg/L AND/OR transferrin saturation ≤20%
* Haemoglobin 110 - 150 g/L

Exclusion Criteria:

* Pregnancy or breast feeding (Female patients of childbearing age will be asked if there is any possibility they may be pregnant. This is standard of care and no pregnancy test will be requested unless there is doubt about this. IV iron is given to many pregnant patients in standard treatment and there is no evidence of harm to mother or foetus).
* Weight < 50kg
* Known allergy to iron therapy
* Haemochromatosis, porphyria cutanea tarda or history of acquired iron overload
* Intravenous iron within previous 6 weeks
* CRP > 50 mg/L
* Serum phosphate < 0.7 mmol/L.
* Active infection
* Current therapy with ESAs
* Uncontrolled atrial fibrillation
* Use of anticoagulants in those under consideration for muscle biopsy
* Unstable angina or heart attack within the last year
* Presence of solid organ cancer
* Known haemoglobinopathy, myelodysplasia, or myeloma
* Patients with peripheral vascular or musculoskeletal disease, who the investigator deems unable to carry out the 6MWT.
* Known severe aortic stenosis and pacemaker in-situ
* History of severe atopy
* Severe liver disease with serum transaminases > x3 upper limit of normal range according to local laboratory values.
* Severe lung disease with FEV1 known to be <50% predicted in last year
* Known heart failure with a left ventricular ejection fraction <45% in last year
* Any other health condition considered by the local Principal Investigator in which IV iron will be contraindicated.
* Insufficient understanding of the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Exercise capacity as measured by 6 minute walk distance (6MWD) | 4 weeks
  An exercise capacity test

SECONDARY OUTCOMES:
Haemoglobin levels | 12 weeks
  Haemoglobin
Iron status | 12 weeks
  Ferritin
Renal function | 12 weeks
  urea,
VO2 peak test (in a sub-set of participants) | 12 weeks
  To assess physical capacity
Isokinetic dynamometry (muscle strength) | 12 weeks
  To assess physical capacity
Functional capacity | 12 weeks
  sit-to-stand 60 to assess lower limb function
KDQOL-36 | 12 weeks
  To assess quality of life by classifying patient general state of health. 1 - Excellent, 2 - Very Good, 3 - Good, 4 - Fair, 5 - Poor.
Skeletal muscle phosphocreatine recovery halftime (PCr t1/2) on MRI spectroscopy (n=40 patients at baseline and 4 weeks) | 12 weeks
  To assess skeletal muscle metabolism
The Work and Social Adjustment Scale (WSAS) | 12 weeks
  To assess quality of life by classifying out more about how participant fatigue impacts on their daily life 0 - Not at all, 1 to 2 - Slightly, 3 to 4 - Definitely, 5 to 6 - markedly and 7 to 8 - Very severely impaired /Cannot work
To assess the impact of iron regulatory genes e.g. HFE, TMPRSS6 etc. on the primary and secondary endpoints of the study (exploratory only) | 12 Weeks
  Patients will be asked if they are willing to provide DNA from a single sample of whole blood to facilitate analysis of up to 90 iron regulatory genes, including HFE and TMPRSS. Iron regulatory gene expression measured by qPCR e.g. Hepcidin, Hemojuvelin, Ferroportin, Trf1 receptor, and iron regulatory proteins-1 & -2.
Iron Status | 12 weeks
  TSAT
Renal Function | 12 weeks
  creatinine
Renal Function | 12 weeks
  estimated glomerular filtration rate to be used to determine renal function

CONTACTS AND LOCATIONS:
Overall Officials: Kate Bramham, Principal Investigator — Kings College Hospital NHS Foundation Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom